CLINICAL TRIAL: NCT00749112
Title: Low Doses of Alemtuzumab and Rituximab in the Treatment of Refractory Autoimmune Cytopenias
Brief Title: Alemtuzumab and Rituximab in the Treatment of Refractory Autoimmune Cytopenias
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: David Gomez-Almaguer, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE08-004
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Anemia, Hemolytic, Autoimmune
Keywords: Idiopathic Thrombocytopenic Purpura; Anemia; Hemolytic; Autoimmune; Alemtuzumab; Rituximab
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Anemia; Hemolysis | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Alemtuzumab, Rituximab

INTERVENTIONS:
Drug: Alemtuzumab, Rituximab — Alemtuzumab 10 mg each 24 hrs subcutaneous for 3 days. Rituximab 100 mg IV every week for 4 weeks.
  Other Names: campath; mabthera

SUMMARY:
The purpose of this study is to determine whether the combination of low doses of alemtuzumab and rituximab are effective in the treatment of patients with autoimmune cytopenias who has failed on steroids, relapsed after steroids withdrawal or required continuous steroids treatment.

DETAILED DESCRIPTION:
Autoimmune cytopenias are a common entities with good responses to steroids therapies as first line, but there is a considerable percentage of patients who relapse, become refractory or dependant on steroids to maintain an acceptable level of hemoglobin or platelets, and the treatment becomes more difficult increasing the secondary effects. The current study evaluates the safety and efficacy of the combination of low doses of alemtuzumab (anti CD52) and Rituximab (anti CD 20) as a second line treatment option for this subset of patients improving the cytopenias without increasing the adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or = 16 years
* Weight: more than 40 Kg
* Autoimmune Hemolytic anemia with clinical and biochemical evidence of hemolysis refractory to treatment, in relapse or steroids dependant
* Idiopathic thrombocytopenic purpura with platelet counts < 50,000, refractory to treatment, in relapse or steroids dependant

Exclusion Criteria:

* Current viral or bacterial infection.
* Positive serology for HIV, HCV, HBV.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate (CR: complete remission, PR: partial remission, relapse rate. | 1, 2, 4 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez-Almaguer, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hopsital Universitario Dr. Jose E. Gonzalez, Centro Universitario contra el Cancer, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Derived] Gomez-Almaguer D, Solano-Genesta M, Tarin-Arzaga L, Herrera-Garza JL, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Jaime-Perez JC. Low-dose rituximab and alemtuzumab combination therapy for patients with steroid-refractory autoimmune cytopenias. Blood. 2010 Dec 2;116(23):4783-5. doi: 10.1182/blood-2010-06-291831. Epub 2010 Sep 14. PMID 20841509